CLINICAL TRIAL: NCT01994239
Title: A Multicenter Randomised Phase II Study Comparing the Efficiency of a HT Concomitant With RT vs RT Alone in the Salvage of Patients With a Detectable PSA After Prostatectomy
Brief Title: Comparison of HT Concomitant With RT vs RT Alone in Patients With a Detectable PSA After Prostatectomy
Acronym: GETUG-AFU22
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UC-0160/1204; 2012-001561-32 (EudraCT Number)
Record Dates: First submitted 2013-10-16; First posted 2013-11-25 (Estimated); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Adenocarcinoma of Prostate
Keywords: Prostate-Specific Antigen; LHRH antagonist; Radiotherapy
MeSH Terms: interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiation (Active Comparator): Pelvic radiotherapy
  * 46 Gy in 23 fractions of 2 Gy.
  * prostate only-boost up to 66 Gy
  Interventions: Radiation: Pelvic Radiotherapy
- Radiation and Degarelix (Experimental): Radiotherapy:
  * 46 Gy in 23 fractions of 2 Gy.
  * prostate only-boost up to 66 Gy
  Associated with hormonal therapy by degarelix:
  * beginning in parallel to radiotherapy for 6 months
  * First dose of 240 mg
  * Maintenance dose of 80 mg
  Interventions: Drug: Degarelix; Radiation: Pelvic Radiotherapy

INTERVENTIONS:
Drug: Degarelix — First dose of 240 mg 5 Maintenance doses of 80 mg every 28 days(+/-3d)
  Other Names: Firmagon
  Arms: Radiation and Degarelix
Radiation: Pelvic Radiotherapy — 46 Gy in 23 fractions Prostate only-boost up to 66 Gy

SUMMARY:
The purpose of this study is to select the best therapeutic strategy in studying the effectiveness of the association of a short duration hormonal therapy and radiotherapy compared with radiotherapy alone, in patients with a detectable PSA after radical prostatectomy.

DETAILED DESCRIPTION:
Study the effectiveness of the association of a short duration hormonal therapy by degarelix (Firmagon ®) and radiotherapy, with radiotherapy alone on survival without events in the treatment of detectable PSA after radical prostatectomy.

122 patients should be included over a period of 2 years. Patients will be treated according to the following scheme:

* Arm A (61 patients) : Pelvic Radiotherapy: 46 Gy and prostate only boost up to 66 Gy
* Arm B (61 patients) : Arm A + hormonal therapy by degarelix during 6 months

ELIGIBILITY:
Inclusion Criteria:

1. Patient with localized prostate adenocarcinoma treated with radical prostatectomy (whatever the initial prognostic stage)
2. R0 or R1
3. pN0 or pNx
4. Post prostatectomy PSA ≥0.2 ng/mL measured between 1 month and 4 months after surgery and increasing to a second test performed between 1 et 8 months after the post prostatectomy dosage
5. PSA ≤2 ng/mL at moment of the randomisation
6. No clinical signs of progressive disease (bone scan or PET scan or abdominal and pelvic scan or MRI): N0, M0
7. Neutrophils ≥1500/mm³; platelet count ≥100 000/mm³
8. Bilirubin ≤ upper limit of normal (ULN); alkaline phosphatase (ALP), aspartate aminotransferase (AST), and Alanine aminotransferase (ALT) ≤1.5 ULN
9. Creatinine <140 µmol/L (or clearance >60 mL/min)
10. Normal fasting glucose
11. Eastern Cooperative Oncology Group (ECOG) ≤1
12. Age >18 years
13. Life expectancy ≥10 years
14. Patients with invasive cancer in complete response for more than five years are eligible
15. Patients who have received the information sheet and signed the informed consent form
16. Patients with a public or a private health insurance coverage

Exclusion Criteria:

1. Prostate cancer histology other than adenocarcinoma
2. Patients pN1, N1 and M1
3. History of pelvic radiotherapy
4. Contraindication to pelvic irradiation (eg, scleroderma, chronic inflammatory bowel disease, etc.)
5. Testosterone ≤0.5 ng/mL
6. History of surgical castration
7. Previous treatment by hormonotherapy
8. Antineoplastic treatment in progress
9. History of another invasive cancer within 5 years before inclusion (with the exception of a basal cell skin carcinoma treated)
10. Known pituitary adenoma
11. Severe hypertension uncontrolled by appropriate treatment (160 mm Hg systolic and/or 90 mm Hg diastolic)
12. Patient with a corrected QT interval (using Fridericia correction) greater than 450 msec
13. Individual deprived of liberty or placed under the authority of a tutor
14. Unable to undergo medical monitoring test for geographical, social or psychological reasons
15. Known hypersensitivity to the treatment in test
16. Administration of an investigational therapeutic within 28 days prior to the screening visit or more if treatment is likely to influence the outcome of this

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-12 (Actual); Primary Completion 2022-03 (Actual); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
The efficacy of the combination of hormonal therapy by degarelix and radiotherapy on event-free survival | 5 years

SECONDARY OUTCOMES:
Survival without biological event | 5 years
  Biochemical recurrence was defined as a PSA > nadir + 0.4 ng / mL confirmed by a second PSA> nadir + 0.4 ng / mL in elevation.
Survival without clinical event | 5 years
  The clinical recurrence will be defined by the discovery of a local recurrence in rectal examination, the appearance of metastases by imaging or biopsy, or clinical manifestation associated with malignant disease without elevated PSA but with histological documentation or imaging.
Survival without metastases | 5 years
Overall survival | 5 years
Acute and late toxicities of the association of hormone therapy with radiotherapy | up to 5 years
  according CTC-AE v4.0
Toxicities of radiotherapy | up to 5 years
  according CTC-AE v4.0
Patient Quality of life | up to 5 years after the end of the radiotherapy
  QLQ-C30, QLQ-PR25 and IPSS
kinetics of testosterone | up to 12 months after the end of the radiotherapy and after biological release

CONTACTS AND LOCATIONS:
Overall Officials: Igor LATORZEFF, Principal Investigator — Clinique Pasteur; Laurent SALOMON, Principal Investigator — CHU Henri Mondor; Paul SARGOS, Principal Investigator — Institut Bergonié; Emmanuel MEYER, Principal Investigator — Centre François Baclesse
Locations (39):
- France (39):
  - Institut de Cancérologie de l'Ouest -Site Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Chu Jean Minjoz, Besançon
  - Institut Bergonié, Bordeaux
  - Centre d'oncologie - Clinique Pasteur, Brest
  - Centre François Baclesse, Caen
  - Centre hospitalier de Chambéry, Chambéry
  - Hôpital Henri Mondor, Créteil
  - Centre d'oncologie et de radiothérapie du Parc, Dijon
  - Centre Georges François Leclerc, Dijon
  - Clinique Sainte-Marguerite, Hyères
  - Chd Vendee, La Roche-sur-Yon
  - Centre Leon Berard, Lyon
  - Clinique Clairval, Marseille
  - CHU La Timone - Hôpital Nord, Marseille
  - Groupe Oncorad Garonne Clinique Du Pont de Chaume, Montauban
  - Ghi Le Raincy / Montfermeil, Montfermeil
  - Centre Azureen de Cancerologie, Mougins
  - Centre Hospitalier Emile Muller, Mulhouse
  - Institut de Cancerologie de Lorraine, Nancy
  - Centre Antoine Lacassagne, Nice
  - Chu Caremeau, Nîmes
  - CHR Orléans La Source, Orléans
  - Hôpital d'Instruction des Armées du Val de Grâce, Paris
  - Hôpital Saint Louis, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de POITIERS, Poitiers
  - Institut Jean Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - Clinique Armoricaine de Radiologie, Saint-Brieuc
  - CHP Saint Grégoire, Saint-Grégoire
  - Institut de Cancérologie de l'Ouest René Gauducheau, Saint-Herblain
  - Clinique Mutualiste de l'Estuaire, Saint-Nazaire
  - Institut de Cancérologie LUCIEN NEUWIRTH, Saint-Priest-en-Jarez
  - Clinique Cote Emeraude, St-Malo
  - Hôpitaux du Léman, Thonon-les-Bains
  - Groupe Oncorad Garonne, Toulouse
  - Centre Marie Curie, Valence
  - GUSTAVE ROUSSY, Cancer Campus, Grand Paris, Villejuif

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.

REFERENCES:
- See also: Site UNICANCER — http://www.unicancer.fr